CLINICAL TRIAL: NCT06677775
Title: A Prospective Clinical Study Based on USTC Diagnostic Model and PSMA/PET-CT for Direct Radical Prostatectomy in Some Patients with First Negative Biopsy
Brief Title: Pathological Positivity Rate in Prostate Cancer Patients with PI-RADS 4 and First Negative Biopsy
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Tao Tao, MD, Associate professor, Associate chief physician, Anhui Provincial Hospital
Other Study IDs: SNOTOB-III
Record Dates: First submitted 2024-11-03; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate biopsy; diagnostic model; mpMRI; prostate specific antigen; PI-ARDS
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this prospective, single-center, single-arm trial was to evaluate the pathologic type of re-treatment based on a clear PI-RADS score of ≥4 with a first negative prostate biopsy, belonging to the high-risk group of the USTC diagnostic model, and PSMA PET/CT positive patients, and to evaluate the diagnostic efficacy of the USTC diagnostic model combined with PSMA PET/CT. At the same time, to explore whether these patients can directly undergo radical prostatectomy without repeated puncture.

Firstly, patients with PI-RADS≥4 scores were screened and the first prostate biopsy was negative. Then USTC diagnostic model was used to evaluate the risk probability of patients suffering from csPCa to determine whether the patients belonged to the high-risk group. Then PSMA/PET-CT was improved for patients in high-risk group to identify the positive lesions of prostate. Finally, for patients with ≥4 PI-RADS and negative prostate aspiration for the first time, Laparoscopic radical prostatectomy (LRP) was performed compared with high-risk groups of USTC diagnostic model and positive PSMA PET/CT. Transperineal targeted prostate biopsy was performed if intraoperative freeze pathology indicated prostate cancer, then LRP was performed; intraoperative freeze pathology indicated benign prostate biopsy, then transperineal prostate biopsy was performed.

DETAILED DESCRIPTION:
Research design This is a prospective, single-center, single-arm, open-label clinical study conducted at the First Affiliated Hospital of the University of Science and Technology of China. Patients with no contraindications to surgery and who meet enrollment criteria will be included in the study. Subsequently, the investigators will recommend that these patients be treated again for PI-RADS≥4, first negative prostate puncture, high-risk group of USTC diagnostic model, and PSMA PET/CT positive patients. Laparoscopic radical prostatectomy (LRP) was directly performed. Transperineal targeted prostate biopsy was performed if intraoperative freeze pathology indicated prostate cancer, then LRP was performed; intraoperative freeze pathology indicated benign prostate biopsy, then transperineal prostate biopsy was performed.

The diagnostic efficacy of USTC diagnostic model combined with PSMA PET/CT was evaluated according to the pathological results of LRP postoperative specimens or prostate biopsy specimens, and whether such patients can directly undergo radical prostatectomy without repeated puncture was also discussed. Before surgery, patients and their families should be fully informed of the surgical risks, the necessity of pathologic confirmation of prostate biopsy, the possibility of benign prostate lesions, and other alternative treatments, including active monitoring, radiotherapy, and focal therapy.

Screening and registration This study consisted of a prostate cancer diagnostic model and a tandem examination of 18F-Prostate-specific membrane antigen 1007 positron emission tomography/computed tomography (18F-PSMA-1007 PET/CT).

For patients with PI-RADS≥4 and negative prostate puncture for the first time, the prostate magnetic resonance score was re-evaluated three months later. For patients with PI-RADS still ≥4, the serum prostate-specific antigen (PSA) test and multi-parameter magnetic resonance imaging (mpMRI) were completed. Prostate-specific antigen density (PSAD) and Prostate Imaging Reporting and Data System version 2.1 (PI-RADS v2.1) score information were obtained. Then through online diagnosis chart (website: https://ustcprostatecancerprediction.shinyapps.io/dynnomapp/) patients with clinically significant probability of the risk of prostate cancer (csPCa). When the csPCa prediction probability is equal to or greater than 0.60, 18F-PSMA-1007 PET/CT is used for further diagnosis. If a patient is still considered to have csPCa after an 18F-PSMA-1007 PET/CT examination, the investigators define this as a positive result. These patients met our study criteria. Notably, patients with a predicted probability of less than 0.60 will no longer receive 18F-PSMA-1007 PET/CT, and patients with a risk probability equal to or greater than 0.60 but negative 18F-PSMA-1007 PET/CT will not meet the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* PI-RADS≥4 scores and the first prostate biopsy was negative
* USTC clinical diagnosis model calculated risk probability value ≥0.6
* Reexamination of PSMA/PET-CT after the first puncture indicated positive prostatic lesions

Exclusion Criteria:

* Life expectancy is less than 15 years
* Multiple metastasis of tumor is possible
* There are serious cardiovascular and cerebrovascular diseases, bleeding tendencies and other surgical or puncture contraindications

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * PI-RADS≥4 scores and the first prostate biopsy was negative
  * USTC clinical diagnosis model calculated risk probability value ≥0.6
  * Reexamination of PSMA/PET-CT after the first puncture indicated positive prostatic lesions
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Reexamination pathologic positive rate of target patients | 2024-2025

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD Ph.D, Study Chair — The First Affiliated Hospital of USTC
Locations (1):
- The First Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No